CLINICAL TRIAL: NCT01226264
Title: Diffusion MRI; Predictive Value for Cervical Uterine Cancer Recurrence.
Acronym: s52647
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, katrijn Michielsen, PhD researcher Radiology, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: s52647
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Uterine Cervical Cancer; Diffusion-weighted MRI; Recurrence
Keywords: Uterine cervical cancer; diffusion-weighted MRI; recurrence
MeSH Terms: conditions — Uterine Cervical Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Diffusion weighted MRI (DW- MRI) — An MRI examination (including diffusion-weighted sequences) belongs to the standard protocol for patients with cervical uterine cancer. The additional burden is therefore restricted to an extra MRI scan during and/or early after therapy.
  MRI is a technique based on magnetic fields and do not require the use of ionizing radiation. Because of the strong magnetic field, a few precautions should be taken. This means that all metal and magnetized objects must be removed from the patient before entering the MRI room. Patients with a pacemaker, a cardiac defibrillator or other implanted conductor/prosthesis are for this reason not eligible for the study.
  During the examination, an intravenous and vaginal contrast medium will be administered. In most cases, patients do not experience any discomfort and the use of these contrast agents is part of the clinical routine.

SUMMARY:
Uterine cervical cancer is the second most common female malignancy. Therapy monitoring is essential to detect early recurrence. Diffusion-weighted magnetic resonance imaging is an emerging MRI imaging technique which has a potential value for the detection of primary and recurrent disease and for the assessment of response to therapy. The purpose of this project is to evaluate the predictive value of DWI during and after therapy in the prediction of recurrence of cervical uterine cancer. It will be considered whether DWI is able to provide early information about the response to therapy. This could enable the identification of less- or non-responsive tumors and in this way therapy can be adapted as soon as possible. Hence the investigators could offer the patient a more efficient treatment scheme and a reduction in toxicity related to the treatment could be established.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cervical uterine cancer are, on a voluntary basis, enrolled in the study. These are patients who either underwent curative chemoradiation (mainly patients with advanced stage cancer) or neoadjuvant chemotherapy (predominantly in patients with early stage cancer) before undergoing surgery.

Exclusion Criteria:

* Patients with known contra-indications for MRI (cardiac pacemakers, cochlear implants, claustrophobic patients) will be excluded from this study. And so are patients with contra-indications to Gadolinium-based contrast agents and patients with a known restricted renal function (GFR < 30 ml/min).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the predictive value of DWI during and after therapy in the prediction of recurrence of cervical uterine cancer. | 2010-2014 continuously
  The purpose of this project is to evaluate the predictive value of DWI during and after therapy in the prediction of recurrence of cervical uterine cancer. It will be considered whether DWI is able to provide early information about the response to therapy.Several studies and a significant experience of our research groups have shown an advantage of DWI for early detection of cancer and evaluation of therapeutic effects [7-10]. This has not yet been demonstrated in patients with cervical uterine cancer. This study aims to expand the scope of the use of DWI.

SECONDARY OUTCOMES:
Reduction in toxicity related to the treatment | 2010-2014
  Nowadays, a large amount of possible treatment schemes for cervical uterine cancer are available but there is an increased need for early and non-invasive treatment follow-up. This could enable the identification of less- or non-responsive tumors and in this way therapy can be adapted as soon as possible. Hence we could offer the patient a more efficient treatment scheme and a reduction in toxicity related to the treatment could be established.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Gasthuisberg, Leuven, Leuven, Belgium